CLINICAL TRIAL: NCT03173742
Title: Bioavailability and Safety of Two Oral Fixed Dose Preparations Containing 18 mg Ivermectin (IVM 18 MG TABLETS, LICONSA S.A., Spain) Versus Reference Dosing (Weight Based) Containing 6 mg Ivermectin (REVECTINA, Abbott Laboratórios do Brasil Ltda, Brazil)
Brief Title: Bioavailability and Safety of Two Oral Fixed Dose Preparations Containing 18 mg Ivermectin (IVM 18 MG TABLETS, LICONSA S.A., Spain) Versus Reference Dosing (Weight Based) Containing 6 mg Ivermectin (REVECTINA®, Abbott Laboratórios do Brasil Ltda, Brazil)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Insud Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MS842-101; 2015-005690-20 (EudraCT Number)
Record Dates: First submitted 2017-05-17; First posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Helminthiasis
MeSH Terms: conditions — Helminthiasis | interventions — Triiodothyronine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- T1, T2, T3 (Experimental): T1: Ivermectin 6 mg (Revectina®) administered according to the SmPC by body weight.
  T2: Ivermectin 18 mg (IVM 18 mg Tablet Liconsa x 1 tablet) T3: Ivermectin 36 mg (IVM 18 mg Tablet Liconsa x 2 tablets)
  Interventions: Drug: T1, T2, T3
- T1, T3, T2 (Experimental): T1: Ivermectin 6 mg (Revectina®) administered according to the SmPC by body weight.
  T2: Ivermectin 18 mg (IVM 18 mg Tablet Liconsa x 1 tablet) T3: Ivermectin 36 mg (IVM 18 mg Tablet Liconsa x 2 tablets)
  Interventions: Drug: T1,T3,T2
- T2,T1,T3 (Experimental): T1: Ivermectin 6 mg (Revectina®) administered according to the SmPC by body weight.
  T2: Ivermectin 18 mg (IVM 18 mg Tablet Liconsa x 1 tablet) T3: Ivermectin 36 mg (IVM 18 mg Tablet Liconsa x 2 tablets)
  Interventions: Drug: T2,T1,T3
- T2,T3,T1 (Experimental): T1: Ivermectin 6 mg (Revectina®) administered according to the SmPC by body weight.
  T2: Ivermectin 18 mg (IVM 18 mg Tablet Liconsa x 1 tablet) T3: Ivermectin 36 mg (IVM 18 mg Tablet Liconsa x 2 tablets)
  Interventions: Drug: T2,T3,T1
- T3,T1,T2 (Experimental): T1: Ivermectin 6 mg (Revectina®) administered according to the SmPC by body weight.
  T2: Ivermectin 18 mg (IVM 18 mg Tablet Liconsa x 1 tablet) T3: Ivermectin 36 mg (IVM 18 mg Tablet Liconsa x 2 tablets)
  Interventions: Drug: T3,T1,T2
- T3,T2,T1 (Experimental): T1: Ivermectin 6 mg (Revectina®) administered according to the SmPC by body weight.
  T2: Ivermectin 18 mg (IVM 18 mg Tablet Liconsa x 1 tablet) T3: Ivermectin 36 mg (IVM 18 mg Tablet Liconsa x 2 tablets)
  Interventions: Drug: T3,T2,T1

INTERVENTIONS:
Drug: T1, T2, T3 — T1: Ivermectin 6 mg (Revectina®) administered according to the SmPC by body weight.
  T2: Ivermectin 18 mg (IVM 18 mg Tablet Liconsa x 1 tablet) T3: Ivermectin 36 mg (IVM 18 mg Tablet Liconsa x 2 tablets)
  Other Names: Treatment 1-2-3
  Arms: T1, T2, T3
Drug: T1,T3,T2 — T1: Ivermectin 6 mg (Revectina®) administered according to the SmPC by body weight.
  T2: Ivermectin 18 mg (IVM 18 mg Tablet Liconsa x 1 tablet) T3: Ivermectin 36 mg (IVM 18 mg Tablet Liconsa x 2 tablets)
  Other Names: Treatment 1-3-2
  Arms: T1, T3, T2
Drug: T2,T1,T3 — T1: Ivermectin 6 mg (Revectina®) administered according to the SmPC by body weight.
  T2: Ivermectin 18 mg (IVM 18 mg Tablet Liconsa x 1 tablet) T3: Ivermectin 36 mg (IVM 18 mg Tablet Liconsa x 2 tablets)
  Other Names: Treatment 2-1-3
  Arms: T2,T1,T3
Drug: T2,T3,T1 — T1: Ivermectin 6 mg (Revectina®) administered according to the SmPC by body weight.
  T2: Ivermectin 18 mg (IVM 18 mg Tablet Liconsa x 1 tablet) T3: Ivermectin 36 mg (IVM 18 mg Tablet Liconsa x 2 tablets)
  Other Names: Treatment 2-3-1
  Arms: T2,T3,T1
Drug: T3,T1,T2 — T1: Ivermectin 6 mg (Revectina®) administered according to the SmPC by body weight.
  T2: Ivermectin 18 mg (IVM 18 mg Tablet Liconsa x 1 tablet) T3: Ivermectin 36 mg (IVM 18 mg Tablet Liconsa x 2 tablets)
  Other Names: Treatment 3-1-2
  Arms: T3,T1,T2
Drug: T3,T2,T1 — T1: Ivermectin 6 mg (Revectina®) administered according to the SmPC by body weight.
  T2: Ivermectin 18 mg (IVM 18 mg Tablet Liconsa x 1 tablet) T3: Ivermectin 36 mg (IVM 18 mg Tablet Liconsa x 2 tablets)
  Other Names: Treatment 3-2-1
  Arms: T3,T2,T1

SUMMARY:
Evaluation of the bioavailability and safety of one oral preparation containing fixed dose 18 mg ivermectin (IVM 18 MG TABLETS, LICONSA S.A., Spain) or two oral preparations containing fixed dose 18 mg ivermectin (IVM 36 MG TABLETS, LICONSA S.A., Spain) vs. reference dosing (weight based) of reference drug containing 6 mg ivermectin (REVECTINA®, Abbott Laboratórios do Brasil Ltda, Brazil) in fasting conditions. A monocentric, open, randomized, single dose, three-period crossover trial in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Caucasian subjects of either gender (male or female) with an age between 18 and 45 years (both inclusive).
2. Medical history and physical examination with no relevant abnormal findings.
3. No evidence of significant disease (organic or psychiatric) based on medical history, physical examination and complementary tests.
4. Laboratory tests (complete hematology, clinical chemistry and urinalysis).
5. Vital signs (systolic and diastolic blood pressure, heart rate and temperature) and electrocardiogram (ECG) record within normal range at screening.
6. Participating female volunteers must use a reliable contraception method not containing hormones. List of accepted contraception method includes barrier methods (i.e. female/male condoms, diaphragms, spermicides), voluntary sterilization (female tubal occlusion) or non-medicated intrauterine devices (IUD) (i.e. inert or copper-releasing). Abstention is not considered a reliable contraception method.
7. For female volunteers only: they must declare that they did not intend to become pregnant in the last month prior to screening and they do not intend to become pregnant during one month following the last study drug administration.
8. Voluntary participation in the study, with written informed consent from the volunteer.
9. The subject agrees to abstain from beverages or food containing methylxanthines (coffee, tea, cola, energy drinks, chocolate etc.), St John's Wort, vitamins, herbal remedies and chewing-gum for 48 hours prior to study drug administration and during each study period.
10. The subject agrees to abstain from beverages or food containing grapefruit for 14 days prior to the first study drug administration and during the study (until last sample from the last period).

Exclusion Criteria:

1. Background of allergy, idiosyncrasy or hypersensitivity to the study drugs or its excipients.
2. Heavy consumer of stimulating drinks (>5 cups of coffee, tea, chocolate or cola drinks per day).
3. Background of alcoholism or drug dependence in the last one year or daily consumption of alcohol > 40 gr/day for men or > 24 gr/day for women.
4. Use of any medication within 15 days prior to taking the study treatment, including over-the-counter medications and medicinal plants (except for the use of paracetamol in short-term symptomatic treatments).
5. Positive serology for hepatitis B, C or HIV.
6. Background or clinical evidence of cardiovascular, respiratory, renal, hepatic, endocrine, gastrointestinal, hematological or neurological disease or other chronic diseases.
7. Smokers or ex-smokers that gave up smoking less than 1 year prior to the study (day 1 of period I)
8. Pregnancy or lactation status for female subjects.
9. Participation in another clinical trial during the 3 months before starting the current trial.
10. Donate blood in the 8 weeks prior to starting the study.
11. Undergone major surgery during the previous 6 months.
12. Clinically significant abnormal ECG with clinical significance in accordance with the CIM's clinical criterion
13. Restrictive vegetarian diet
14. Positive results to the breath alcohol test at screening or at Day -1
15. Positive results to the drug abuse checks (urine test for: amphetamines, cannabinoids, opiates, benzodiazepines and cocaine) at screening or at admission on Day -1
16. Epidemiological risk of being infected by Loa loa or other filariases, defined as those who have lived or have travelled to any of the following countries: Angola, Cameroon, Central Africa Republic, Chad, Congo, Democratic Republic of the Congo, Equatorial Guinea, Ethiopia, Gabon, Nigeria and Sudan.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Primary endpoint evaluated will be the PK parameters that define bioavailability in extent Ln [AUC0t] | up to day 7
  For group 3
Primary endpoint evaluated will be the PK parameters that define bioavailability in extent in rate: Ln [Cmax] for each treatment in healthy volunteers with high weight (Group 3), calculated by means of a non-compartmental analysis. | up to day 7
  For group 3

SECONDARY OUTCOMES:
Relative bioavailability for each treatment and for groups 1 and 2 will be evaluated with the PK parameters that define bioavailability in extent Ln [AUC0t] | up to day 7
  for group 1 and 2
Relative bioavailability for each treatment and for groups 1 and 2 will be evaluated with the PK parameters that define bioavailability in extent in rate: Ln [Cmax] | up to day 7
  for group 1 and 2
AUC0t (for non-compartmental analysis) | up to day 7
  PK profile for each treatment and each study group will be evaluated by means of a compartmental and non-compartmental analysis
AUC0∞ (for non-compartimental analysis) | up to day 7
  PK profile for each treatment and each study group will be evaluated by means of a compartmental and non-compartmental analysis
%AUC extra (residual area) (for non-compartimental analysis) | up to day 7
  PK profile for each treatment and each study group will be evaluated by means of a compartmental and non-compartmental analysis
tmax (for non-compartimental analysis) | up to day 7
  PK profile for each treatment and each study group will be evaluated by means of a compartmental and non-compartmental analysis
tlag (for non-compartimental analysis) | up to day 7
  PK profile for each treatment and each study group will be evaluated by means of a compartmental and non-compartmental analysis
Cl/F (for non-compartimental analysis) | up to day 7
  PK profile for each treatment and each study group will be evaluated by means of a compartmental and non-compartmental analysis
V/F (for non-compartimental analysis) | up to day 7
  PK profile for each treatment and each study group will be evaluated by means of a compartmental and non-compartmental analysis
t1/2 (for non-compartimental analysis) | up to day 7
  PK profile for each treatment and each study group will be evaluated by means of a compartmental and non-compartmental analysis
Ke (for non-compartimental analysis) | up to day 7
  PK profile for each treatment and each study group will be evaluated by means of a compartmental and non-compartmental analysis
MRT (for non-compartimental analysis) | up to day 7
  PK profile for each treatment and each study group will be evaluated by means of a compartmental and non-compartmental analysis
Cmax (for non-compartimental analysis) | up to day 7
  PK profile for each treatment and each study group will be evaluated by means of a compartmental and non-compartmental analysis
tlag (for compartimental analysis) | up to day 7
  PK profile for each treatment and each study group will be evaluated by means of a compartmental and non-compartmental analysis
ka (for compartimental analysis) | D7
  PK profile for each treatment and each study group will be evaluated by means of a compartmental and non-compartmental analysis
Cl/F(for compartimental analysis) | up to day 7
  PK profile for each treatment and each study group will be evaluated by means of a compartmental and non-compartmental analysis
V/F (for compartimental analysis) | up to day 7
  PK profile for each treatment and each study group will be evaluated by means of a compartmental and non-compartmental analysis
vital signs | up to week 6
  To asses safety and tolerability of the treatments
laboratory analysis | up to week 6
  To asses safety and tolerability of the treatments
Incidence of adverse events. | up to week 6
  To asses safety and tolerability of the treatments
ECG | up to week 6
  To asses safety and tolerability of the treatments

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Munoz J, Ballester MR, Antonijoan RM, Gich I, Rodriguez M, Colli E, Gold S, Krolewiecki AJ. Safety and pharmacokinetic profile of fixed-dose ivermectin with an innovative 18mg tablet in healthy adult volunteers. PLoS Negl Trop Dis. 2018 Jan 18;12(1):e0006020. doi: 10.1371/journal.pntd.0006020. eCollection 2018 Jan. PMID 29346388